CLINICAL TRIAL: NCT06539806
Title: Clinical Study Evaluating the Effect of Losartan on Response Rate in Both Metastatic and Locally Advanced Pancreatic Cancer Patients
Brief Title: Clinical Study Evaluating the Effect of Losartan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Abd El- Rafea Abdo, Assistant lecturer of Clinical Pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mona Abd El-Rafea Mohamed
Record Dates: First submitted 2024-07-18; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Losartan; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (locally advanced PC patients): (Active Comparator): Including three subset groups (A, B and C)
  •Group I- A(control group): Fifteen hypertensive patients treated with antihypertensive agent except ARBS and ACEI with locally advanced PC on Folfirinox.
  • Group I -B (are not treated with ARBs or ACEI prior PC diagnosis): Fifteen hypertensive patients with locally advanced PC and are not treated with ARBs or ACEI before PC diagnosis on the same chemotherapy treatment protocol as the control group in addition to losartan 50 mg once daily for one year after PC diagnosis.
  • Group I-C (losartan was used for treatment of hypertension before and after PC diagnosis):Fifteen hypertensive patients with locally advanced PC and were treated with losartan one year before PC diagnosis on the same chemotherapy treatment protocol as the control group in addition to losartan 50 mg once daily for one year after PC diagnosis and the dose will be titrated up according to the patient's response.
  Interventions: Drug: Losartan 50mg Tab
- Group II (metastatic PC patients): (Active Comparator): including three subset groups (A, B and C):
  • Group II-A (control group): Fifteen hypertensive patients treated with antihypertensive agent except ARBS and ACEI with metastatic PC on Gemcitabine hydrochloride 1 gm. vial taken as 1000 mg/m2 IV over 30 min weekly for 7 weeks.
  • Group II-B (are not treated with ARBs or ACEI prior diagnosis): Fifteen hypertensive patients with metastatic PC and are not treated with ARBs or ACEI before PC diagnosis on the same chemotherapy treatment protocol as the control group in addition to Losartan 50 mg once daily for one year after PC diagnosis.
  • Group II-C (losartan was used for treatment of hypertension before and after PC diagnosis): Fifteen hypertensive patients with metastatic PC and were treated with losartan one year before PC diagnosis and on the same chemotherapy treatment protocol as the control group in addition to Losartan 50 mg once daily for one year after PC diagnosis
  Interventions: Drug: Losartan 50mg Tab

INTERVENTIONS:
Drug: Losartan 50mg Tab — The efficacy of losartan on response rate in both metastatic and locally advanced pancreatic cancer patients
  Other Names: Gemcitabine hydrochloride

SUMMARY:
The pancreas is two organs packaged into one. The islets of Langerhans serve critical endocrine functions, and the exocrine portion is a major source of enzymes that are essential for digestion.

Pancreatic cancer (PC) is more commonly referred to as pancreatic infiltrating ductal adenocarcinoma in addition to being the second leading cause of cancer death in the United States, after lung cancer in 2020.

Whereas pancreatic cancer is the seventh cause of death from cancer in Asia in 2020. Although it is substantially less common than the other malignancies, pancreatic carcinoma is near the top of the list of killers because it is a highly aggressive carry.

DETAILED DESCRIPTION:
Pancreatic cancer has multi step carcinogenesis, starting from Pancreatic Intra-ductal Neoplasia and ends with an invasive neoplastic lesion.Pancreatic cancer is most frequent in elder people; the risk of developing pancreatic cancer goes up as people age.

It is frequently found at an advanced stage, which contributes to five-year survival rates of 2-9%, ranking firmly the pancreatic cancer among all cancer sites in terms of prognostic outcomes for patients. In addition, it has a high trend to show nodal metastasis, hepatic, bone, or pulmonary metastasis.

Epidemiological data shows that pancreatic cancer is not very common but obvious it is one of the most neoplastic death-cause in the world.The Renin angiotensin system (RAS) is an important regulator of the cardiovascular system that was identified. in this system, angiotensinogen is converted to angiotensin (Ang) I and then to Ang II by renin and angiotensin-converting enzyme (ACE), respectively.

The Ang II activates the angiotensin type 1 receptor (AT1R). It has been suggested that RAS components are involved in the evolution of various cancers and tissues, like prostate, skin, and pancreatic cancer. In the pancreas, they are considered to mediate growth and lead to carcinogenesis.

High concentrations of Ang II have been reported together with up-regulated levels of AT1R in human with pancreatic cancer and malignant pancreatic tissues.

AT1R is known to activate phosphatidylinositol-specific-phosphodiesterase C enzyme after being activated by Ang II to produce phosphate inositol and 2-acylglycerol, which causes the entry of Ca2+ into cells, hence, activating protein kinase C and mitogen-activated protein kinase (MAPK).

MAPK has an important role in cell proliferation. Moreover, studies show that Ang II induces Vascular endothelial growth factor (VEGF) expression which is the main growth factor involved in angiogenesis.

Several studies have reported that RAS can increase the risk of metastasis in various cancers. Building upon these findings, RAS blockers may be expected to be beneficial in pancreatic cancer treatment.

Losartan is a RAS inhibitor currently well-known to decrease blood pressure. 10 It is demonstrated in several studies that Losartan can inhibit the effect of Ang II on cell proliferation and angiogenesis. In PC, it's suggested that Losartan increases drug delivery to the tumor, thus improving the chemotherapy effect.

Furthermore it increase the efficacy of Nano-therapeutics in pancreatic cancer of mice through enhancing both interstitial and trans-vascular transport. In another study it was found that Losartan raised DNA incorporation of Gemcitabine and enhanced its efficacy.

Studies

Over the past two decades have provided important information on the potential therapeutic use of RAS blocker drugs in cancer.Extensive preclinical data support the potential use of angiotensin II receptor blockers (ARBs) as anti-neoplastic agents in pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* Male and female pancreatic cancer patients aged ≥ 50 years old.
* Hypertensive patient with BP ≥ 140/90 mm Hg.
* Histologically confirmed metastatic pancreatic adenocarcinoma; or locally advanced pancreatic cancer patients.
* All included patients must sign an informed consent

Exclusion Criteria:

* Patients with serious concomitant systemic disorders as significant cardiac, renal, hepatic, or pulmonary morbidity.
* Pregnant or lactating women and women of childbearing potential.
* Patients received prior systemic fluoropyrimidine therapy within the past 10 years.
* Prior un-anticipated severe reaction to fluoropyrimidine therapy, or known hypersensitivity to 5-fluorouracil, irinotecan, oxaliplatin, losartan, or any monoclonal antibody.
* Patients with an active, known, or suspected autoimmune disease such as psoriasis.
* Patients with a known positive test for hepatitis B virus surface antigen (HBV s Ag) or hepatitis C virus (HCV antibody) and patients with a known history of testing positive for (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Patients received a live vaccine or live attenuated vaccines as intranasal influenza vaccines within 30 days of the planned start of study therapy.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
the patient response rate | one year
  the patient response rate which will be measured using response evaluation criteria in solid tumors (RECIT 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Osama Mohamed Hassan, Professor, Study Director — Clinical Pharmacy Department Faculty of Pharmacy, Tanta University; Sahar Mohamed El-Ghobashy, Professor, Study Director — Clinical Pharmacy Department Faculty of Pharmacy, Tanta University; Mohamed Abdel Hamid Mohamed, Professor, Study Chair — Clinical Oncology Faculty of Medicine, Tanta University
Locations (1):
- Tanta University Hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided